CLINICAL TRIAL: NCT04784975
Title: Bone Health and Gut Microbiome in Persons With Preclinical and Clinical Type 1 Diabetes
Brief Title: Bone Health and Microbiome in Persons With Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Anna Neyman, Assistant Professor of Clinical Pediatrics, Indiana University
Other Study IDs: BONE
Record Dates: First submitted 2021-02-26; First posted 2021-03-05 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Type1diabetes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Preclinical Type 1 Diabetes: Adolescents and young adults with preclinical diabetes (having at least 2 positive diabetes autoantibodies but who do not meet criteria for clinical diagnosis of type 1 diabetes).
  There is no intervention. Each group will complete a bone health assessment, a microbiome assessment and a glycemic assessment with the goal of better understanding the association between these different variables and bone health.
  Interventions: Other: No intervention
- New Onset Type 1 Diabetes: Adolescents and young adults with a diagnosis of clinical type 1 diabetes. There is no intervention. Each group will complete a bone health assessment, a microbiome assessment and a glycemic assessment with the goal of better understanding the association between these different variables and bone health.
  Interventions: Other: No intervention
- Long standing Type 1 Diabetes: Adolescents and young adults with type 1 diabetes for at least 2 years. There is no intervention. Each group will complete a bone health assessment, a microbiome assessment and a glycemic assessment with the goal of better understanding the association between these different variables and bone health.
  Interventions: Other: No intervention
- Control: Adolescents and young adults without any evidence of diabetes or hyperglycemia. There is no intervention. Each group will complete a bone health assessment, a microbiome assessment and a glycemic assessment with the goal of better understanding the association between these different variables and bone health.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
It is well-established that persons with type 1 diabetes (T1D) are at an increased risk for morbidity and mortality related to bone fracture due to poor bone health, however we do not fully understand the mechanism behind the increased fracture risk. We are examining bone health and the microbiome in adolescents and young adults with type 1 diabetes to better understand the reasons behind this increased risk.

DETAILED DESCRIPTION:
This pilot study aims to look at measures of bone health, the gut microbiome and measures of glycemia/glycemic variability in those with preclinical and clinical diabetes. Our primary and secondary outcomes are to characterize these variables, with our long term objectives to better understand the natural history of bone health in T1D, help characterize the etiology of worse bone health in those with T1D, and try to identify potential time periods for intervention.

ELIGIBILITY:
Inclusion Criteria:

- Willing and able to comply with study protocol

For participants with type 1 diabetes (T1D):

- T1D diagnosed clinically by an endocrinologist as documented in medical records.

Exclusion Criteria:

* use of oral or parenteral antibiotics within 3 months
* use of probiotics/prebiotics/synbiotics within 3 months of enrollment; persons who eat yogurt will be asked to stop for 30 days prior to stool collection
* use of medications that will affect bone, including glucocorticoids, bisphosphonates
* chronic medications (other than insulin for those with T1D or a stable dose of thyroid hormone)
* uncontrolled chronic gastrointestinal disease including celiac disease (persons with T1D will be screened for celiac disease with a Tissue Transglutaminase Antibody (tTG)/Immunoglobulin A (IgA) if not done in prior 2 years)
* known genetic syndrome that predisposes the participant to fracture (such as osteogenesis imperfect) or skeletal dysplasia that would affect skeletal assessment (such as hypochondroplasia)
* pregnancy
* Any other condition that in the opinion of the investigator would jeopardize the safety or rights of the subject participating in the study or would make it unlikely the subject could complete the study

Additional Exclusion Criteria for Healthy Controls:

* Presence of any diabetes autoantibody
* Presence of any type of diabetes or hyperglycemia (HbA1c≥5.7%)

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Type 1 Diabetes
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2021-04-23 (Actual); Primary Completion 2022-09-23 (Actual); Study Completion 2022-09-23 (Actual)

PRIMARY OUTCOMES:
High-resolution peripheral quantitative computed tomography (HRpQCT) strength of cortical and trabecular bone. | Through study completion, which is within 12 weeks of visit 1
  Our primary outcome is HRpQCT strength of cortical and trabecular bone.

SECONDARY OUTCOMES:
Dual-energy x-ray absorptiometry (DXA) | Through study completion, which is within 12 weeks of visit 1
  Lumbar spine, hip, and total body less head by DXA
Microbiome | Through study completion, which is within 12 weeks of visit 1
  Gut microbiome profile
Glycemia | Through study completion, which is within 12 weeks of visit 1
  Serum Hemoglobin A1C (HbA1c) and Time in Range using a continuous glucose monitor (CGM)

CONTACTS AND LOCATIONS:
Locations (1):
- IUSM, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No